CLINICAL TRIAL: NCT06326697
Title: A Randomized, Single Oral Dose, Open Label, Two Sequence, Two Treatment, Four Periods, Full Replicate Crossover Study to Determine the Bioequivalence of Azacitidine 300 mg Film- Coated Tablets Versus Onureg® 300 mg Film-Coated Tablets for Adult Patients With Acute Myeloid Leukaemia (AML) Under Fasting Conditions
Brief Title: Bioequivalence of Azacitidine 300 mg Film-Coated Tablets in Adult Patients With Acute Myeloid Leukaemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HIK-AZA-2023-01
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Product: Azacitidine 300 mg Film coated tablets (Experimental): Single oral dose of Azacitidine 300 mg Film coated tablets
  Interventions: Drug: Azacitidine
- Reference Product: Onureg® 300 mg Film Coated Tablets (Active Comparator): Single oral dose of Onureg® 300 mg Film Coated Tablets
  Interventions: Drug: Onureg

INTERVENTIONS:
Drug: Azacitidine — Azacitidine 300 mg Film coated tablets
  Arms: Test Product: Azacitidine 300 mg Film coated tablets
Drug: Onureg — Azacitidine 300 mg Film coated tablets
  Arms: Reference Product: Onureg® 300 mg Film Coated Tablets

SUMMARY:
A Randomized, Single Oral Dose, Open Label, Two Treatment, Crossover study to investigate the bioequivalence of the Test Product Azacitidine 300 mg Film coated tablets relative to Reference Product Onureg® 300 mg Film Coated Tablets in adult patients with AML under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Patients age ≥ 18 years of age at the time of signing the informed consent document.
2. Patients with documented diagnosis of AML according to the 2022 updates of the World Health Organization (WHO) classification of myeloid neoplasms and acute leukaemia.
3. Patients with acute myeloid leukemia who achieved first complete remission or complete remission with incomplete blood count recovery following intensive induction chemotherapy and are not able to complete intensive curative therapy. The definitions of response criteria for CR or CRi are primarily those defined by the 2022 report from the European Leukemia Net (ELN) on AML as below: CR defined as bone marrow blasts <5%; absence of circulating blasts; absence of extramedullary disease; ANC ≥ 1.0 × 10^9/L (1,000/µL); platelet count ≥ 100 × 10^9/L(100 000/µL).

   CRi defined as all CR criteria, except for residual neutropenia < 1.0 × 10^9/L (1,000/µL) or thrombocytopenia < 100 × 10^9/L (100 000/µL).
4. Patients who don't have a known or suspected hypersensitivity to Azacitidine or any other ingredient used in the manufacturing of Azacitidine.
5. Patients who are physically able for appropriate pharmacokinetics sampling according to principal investigator evaluation.
6. Patients who have a haematological profile appropriate for receiving Azacitidine 300 mg dose for 4 consecutive days as per the principal investigator assessment.
7. Patients who understand and voluntarily sign a written informed consent document prior to any study related assessments/procedures are conducted.
8. Patient is capable of consent.
9. Females of childbearing potential may participate, providing the subject meets the following conditions: Negative serum pregnancy test at screening (sensitivity of at least 25 mIU/mL), and willing to use effective contraception during and up to 6 months after study.
10. Male patients must be willing to use effective contraception during and up to 3 months after the study.

Exclusion Criteria:

1. Patients with history of drug or alcohol abuse.
2. Female patients who are pregnant or nursing (lactating).
3. Patients with medical condition, laboratory abnormality, or psychiatric illness that, in the opinion of the investigator, might interfere with subject safety, compliance or evaluation of the condition of the study.
4. Patients with positive blood screen for HIV, Hepatitis B (HbsAG) or Hepatitis C (HCV) virus.
5. Patients with experience in any investigational drug in a clinical study within 6 months prior to study Day 1.
6. Patients has a difficulty fasting or consuming standard meals.
7. Patients has history of difficulties in swallowing or any gastrointestinal disease which could affect the drug absorption.
8. Patients does not agree to not be engaged in strenuous exercise at least one day prior to study drug administration until donating the last sample of the study.
9. Patients does not agree to not consuming any beverages or food containing grapefruit for at least two weeks prior to first study drug administration until donating the last sample of the study.
10. Patients does not agree to not consuming any beverages or food containing methyl-xanthines e.g., caffeine (coffee, tea, cola, energy drinks, chocolate etc.) at least 48 hours prior to first study drug administration until donating the last sample of the study.
11. Patients does not agree to not consuming any alcohol containing beverages and food at least 48 hours prior to first study drug administration until donating the last sample of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-08-17 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Cmax | 5 hours
  Maximum measured plasma concentration over the time span specified
AUC0-t | 5 hours
  The area under the plasma concentration versus time curve, from time (0) to the last measurable concentration (t), as calculated by the linear trapezoidal method.

SECONDARY OUTCOMES:
AUC0-∞ | 5 hours
  The area under the plasma concentration versus time curve from time (0) to infinity.
Kel | 5 hours
  Apparent first-order elimination or terminal rate constant
Tmax | 5 hours
  Time of the maximum measured plasma concentration.
T1/2el | 5 hours
  The elimination or terminal half-life.
Adverse Events (AEs) | Day 4
  Adverse Events (AEs)
Change in clinical safety labs | Day 4
  Descriptive Change in clinical safety labs

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No